CLINICAL TRIAL: NCT00165659
Title: A Multi-Center, Randomized, Double-Blind, Parallel Group Study With 3 Groups Receiving Placebo, 5 mg of E2020 and 10 mg of E2020
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2020-J081-231
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

INTERVENTIONS:
Drug: DONEPEZIL HYDROCHLORIDE

SUMMARY:
To evaluate the dose-response efficacy of E2020 (5 mg/day and 10 mg/day) versus placebo and verify superiority of E2020 to placebo in patients with severe AD using CIBIC-plus* and SIB** as the primary efficacy measures. Safety of E2020 will also be evaluated.

(*for overall evalution of clinical symtoms) (**for cognitive function test)

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnostics of Alzheimer's disease (AD) according to DSM-IV.
* Patients with modified Hachinski Ischemic scale score of ≦6.
* FAST score of ≧6 at baseline (4 weeks before starting study treatment).
* MMSE score between 1 and 12 at baseline (4 weeks before starting study treatment).
* Imaging diagnostics (CT, MRI, etc., within 24 months consistent with the diagnosis of AD without any other comorbid pathologies found. If a significant change in clinical status suggesting other types of dementia (except AD) is suspected between the final image diagnosis and the time of starting observation, the scan test should be repeated.
* Patients who can comply with the requirements on concomitant drugs/therapies from the baseline phase or before.
* Patients aged 50 years or older.
* Outpatients. Even in the case of an outpatient or a patient attending on the outpatient-visit basis from a nursing home facility, the caregiver must be a constant and reliable informant with minimum of 3 days per week direct contact with the patient (for at least 4 hours per day on waking hours). This contact is necessary to ensure accurate reporting of the patient's behavior and his/her ability to perform ADLs.
* Patients who are expected to complete all procedures scheduled during the Screening and Baseline visit and who have a reliable caregiver or family member who agrees to accompany the patient to all clinic visits, provide information about the patient as required by the protocol, and ensure compliance with the treatment schedule.
* Patients who can swallow tablets without pulverization.
* Patients who are ambulatory at least aided (walker) and have vision and hearing necessary for compliance with testing procedures (eyeglasses and/or hearing aid permissible).
* Patients whose representatives can sign the written informed consent.

Exclusion Criteria:

* Patients with dementia other than AD.

  1. Patient whose imaging test shows "circumscribed cerebral lesion or multiple infarcts" which is suspected to be the responsible cause of dementia (mixed-type dementia)
  2. Patients with other types of dementia
* Patients with a current DSM-IV diagnosis of major depressive disorder or any current serious psychiatric diagnosis othe than AD.
* Patients without a reliable caregiver.
* Patients who are expected to enter a nursing home facility within 6 months after starting study treatment (excluding a transient entry).
* Patients with active or clinically significant conditions affecting absorption, distribution or metabolism of study drugs (e.g., inflammatory bowel disease, gastric or duodenal ulcers, or severe lactose intolerance).
* Patients with a known hypersensitivity to a component of donepezil hydrochloride preparation or piperidine derivatives.
* Patients complicated with a severe gastrointestinal, hepatic, renal, endocrine, or cardiovascular system disease (e.g., sick sinus syndrome, intraarterial and supraventricular conduction disorder, etc.).
* Patients with a history of severe bronchial asthma or obstructive pulmonary disease.
* Patients with a severe extrapyramidal disease (Parkinson's disease, Parkinson's syndrome, etc.).
* Patients with diabetes mellitus with uncontrolled blood glucose levels (HbAlc of ≧10%).
* Hypertension patients with uncontrolled blood pressure (diastolic blood pressure of ≧95 mmHg).
* Patients with uncontrolled thyroid dysfunction.
* Patients with a history of seizure or convulsion within the previous 3 months (obtaining informed consent).
* Patients with a known or suspected history of alcohoism or drug dependence within the recent 10 years.
* Patients with malignant tumors.
* Women of pregnant, possibly pregnant, or lactating.
* Patients who have participated in another clinical study within the recent 3 months (before giving consent).
* Any other patients who are judged to be ineligible for study entry by the investigator or subinvestigator.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2002-11; Primary Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Primary Outcomes: Efficacy:
CIBIC plus*, SIB**
(*for overall evalution of clinical symtoms)
(**for cognitive function test)
Safety:
Adverse event, adverse drug reaction, vital sign, clinical laboratory parameter, electrocardiogram

SECONDARY OUTCOMES:
Efficacy
Behave-AD, ADCS-ADL-sev

CONTACTS AND LOCATIONS:
Overall Officials: Itaru Arimoto, Study Director — Eisai Co., Ltd - Development Clinical Research Dept., Clinical Research Center
Locations (54):
- Japan (54):
  - Chita, Aichi-ken
  - Nagoya, Aichi-ken
  - Toyohashi, Aichi-ken
  - Akita, Akita
  - Daisen, Akita
  - Kashiwa, Chiba
  - Fukui-shi, Fukui
  - Fukuoka, Fukuoka
  - Kitakyushu, Fukuoka
  - Fukushima, Fukushima
  - Kōriyama, Fukushima
  - Fujioka, Gunma
  - Numata, Gunma
  - Hiroshima, Hiroshima
  - Ōtake, Hiroshima
  - Asahikawa, Hokkaido-prefecture
  - Aio, Hyōgo
  - Asago, Hyōgo
  - Kako, Hyōgo
  - Kobe, Hyōgo
  - Tsuchiura, Ibaraki
  - Tsukuba, Ibaraki
  - Kanazawa, Ishikawa-ken
  - Kawasaki, Kanagawa
  - Sagamihara, Kanagawa
  - Kochi, Kochi
  - Kyoto, Kyoto
  - Nagasaki, Nagasaki
  - Sasebo, Nagasaki
  - Kashihara, Nara
  - Jōetsu, Niigata
  - Kashiwazaki, Niigata
  - Tsukubo, Okayama-ken
  - Moriguchi, Osaka
  - Neyagawa, Osaka
  - Osaka, Osaka
  - Suita, Osaka
  - Takatsuki, Osaka
  - Saitama, Saitama
  - Izumo, Shimane
  - Shizuoka, Shizuoka
  - Kawachi, Tochigi
  - Shimotsuga, Tochigi
  - Chiyoda-ku, Tokyo
  - Hachiōji, Tokyo
  - Higashimurayama, Tokyo
  - Itabashi-ku, Tokyo
  - Kodaira, Tokyo
  - Machida, Tokyo
  - Shinjuku-ku, Tokyo
  - Nanto, Toyama
  - Gobō, Wakayama
  - Wakayama, Wakayama
  - Hōfu, Yamaguchi